CLINICAL TRIAL: NCT04379011
Title: Brivaracetam to Reduce Neuropathic Pain in Chronic SCI: A Pilot Clinical Trial
Brief Title: Brivaracetam to Reduce Neuropathic Pain in Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Morse
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — brivaracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brivaracetam Group (Experimental): Participants in this arm will receive the investigational drug, Brivaracetam.
  Interventions: Drug: Brivaracetam
- Control Group (Placebo Comparator): Participants in this arm will receive a placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Brivaracetam — Escalating brivaracetam dose to 150 mg twice daily for 3 months
  Other Names: Briviact
  Arms: Brivaracetam Group
Other: Placebo — Placebo twice daily for 3 months
  Arms: Control Group

SUMMARY:
Spinal cord injury (SCI) is associated with severe neuropathic pain that is often refractory to all pharmacological intervention. Preliminary data suggest brivarecetum is a mechanism-based pharmacological intervention for neuropathic pain in SCI. This randomized, placebo-controlled pilot clinical trial will assess feasibility of a 3-month treatment course with brivarecetum.

DETAILED DESCRIPTION:
The investigations will assess changes in pain intensity and periaqueductal gray hyperactivity. Baseline periaqueductal gray hyperactivity and microRNA levels will be measured as potential biomarkers of response to treatment. These preliminary findings will be used to design larger clinical trials to establish efficacy of brivarecetum to treat neuropathic pain in SCI.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (SCI)
* Participants must have completed inpatient rehabilitation and are living in the community
* Participant who have severe below-level neuropathic pain (daily average 9/10 or 10/10)
* Participants must have tried and failed to achieve adequate pain relief with the use of other drugs (i.e treatment failed to decrease their pain below a level of 9) and can continue to take spasmolytics, pregabalin, gabapentin, and opioids in unchanged dosing throughout the trial

Exclusion Criteria:

* Pprogressive myelopathy secondary to posttraumatic cord tethering
* Syringomyelia
* Brain injury limiting the ability to follow directions
* Pregnancy or lactation
* Epilepsy
* Impaired liver or renal function
* Contraindications to brivaracetam or pyrrolidine derivatives including allergy, or contraindications to MRI including retained bullet fragments, noncompatible metal implants, and implanted devices such as baclofen pumps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morse, DO, Study Director — University of Minnesota; Scott Falci, MD, Principal Investigator — Swedish Hospital
Locations (2):
- United States (2):
  - Swedish Hospital, Englewood, Colorado
  - University of Minnesota School of Medicine, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Brivaracetam Group
Started | 12 | 12
Completed | 9 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Brivaracetam Group | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (7.9) | 43.5 (12.5) | 47.10 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 10 | 18
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory, Worst Pain
Description: The Brief Pain Inventory (BPI) contains 11 numeric rating scales that measure pain intensity and the effect of the pain on a participant's ability to function during various activities of daily living. Each of the 11 scales is rated from 0 (no pain/does not interfere) to 10 (severe pain/completely interferes). Total scores range from 0-110, with higher scores indicating greater pain and interference on daily activities.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on scale | 8.9 (1) | 9.7 (0.8)

2. Primary Outcome: Brief Pain Inventory, Worst Pain
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on scale | 8.1 (1.6) | 7.8 (1.7)

3. Primary Outcome: Brief Pain Inventory, Least Pain
Description: as for outcome 1
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on scale | 5.1 (3.3) | 4.8 (3.2)

4. Primary Outcome: Brief Pain Inventory, Least Pain
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on scale | 5.6 (2.4) | 4.7 (3.4)

5. Primary Outcome: Brief Pain Inventory, Average Pain
Description: as for outcome 1
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on scale | 6.7 (1.8) | 7.5 (1.6)

6. Primary Outcome: Brief Pain Inventory, Average Pain
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on scale | 6.4 (1.9) | 7 (1.8)

7. Primary Outcome: Satisfaction With Life Scale (SWLS)
Description: The satisfaction with life scale contains 5 items designed to measure global cognitive judgments of life satisfaction. Each of the 5 items is rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). Total scores range from 5 to 35, with higher scores indicating greater satisfaction with life.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on a scale | 17.9 (7) | 20.2 (5.6)

8. Primary Outcome: Satisfaction With Life Scale (SWLS)
Description: as for outcome 7
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Brivaracetam Group
Number analyzed (Participants) | 8 | 6
score on a scale | 18.3 (8.4) | 19.8 (8.1)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Control Group | Brivaracetam Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/11
Other Adverse Events (participants affected / at risk) | 8/9 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=9) | Brivaracetam Group (N=11)
hospitalization due to nausea and vomiting (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=9) | Brivaracetam Group (N=11)
gastrointestinal symptoms (Gastrointestinal disorders) | 0 (0) | 5 (9)
neurological symptoms (Nervous system disorders) | 3 (3) | 5 (6)
fatigue (General disorders) | 2 (2) | 5 (5)
psychological symptoms (General disorders) | 2 (2) | 3 (3)
vasomotor symptoms (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The protocol did not allow for assessment of pain scores prior to or after the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT04379011/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT04379011/ICF_001.pdf